CLINICAL TRIAL: NCT00354367
Title: A Phase IIIB Multicenter, Open Label, Randomized Clinical Trial Evaluating Efficacy of Certolizumab Pegol, a PEGylated Fab Fragment of Humanized Antibody to Tumor Necrosis Factor (TNF) in Crohn's Disease Patients With Draining Fistulas.
Brief Title: Evaluate Efficacy of Certolizumab in Crohn's Patients With Draining Fistulas
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C87058
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Certolizumab pegol; Fistula
MeSH Terms: conditions — Crohn Disease; Fistula | interventions — Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab pegol

SUMMARY:
To investigate the clinical efficacy of certolizumab pegol for fistula closure in Crohn's disease subjects with active draining fistulas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single or multiple fistulas, including perianal and enterocutaneous fistulas for at least 3 months as a complication of Crohn's disease

Exclusion Criteria:

* Symptomatic obstructive intestinal strictures, bowel resection, proctocolectomy or total colectomy, abscesses present at screening, current total parenteral nutrition, short bowel syndrome.
* All the concomitant diseases or pathological conditions that could interfere with Crohn's disease assessment or to be harmful for the well being of the patient.
* Previous clinical trials and previous biological therapy that could interfere with the results in the present clinical trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Investigation of Clinical efficacy of certolizumab pegol for fistula closure, as measured by the proportion of patients with fistula improvement after 16 weeks of treatment.

SECONDARY OUTCOMES:
Investigation of Clinical efficacy of certolizumab pegol for maintenance of fistula closure.

CONTACTS AND LOCATIONS:
Overall Officials: Krassimir Mitchev, MD, Study Director — UCB / Global Medical Affairs